CLINICAL TRIAL: NCT04755140
Title: Evaluation and Clinical Impact of Serum and Blood Metal Ion Levels in Patients With an Endoprosthesis
Brief Title: Endoprosthesis Metal Toxicity Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-008408; R01AG060920 (NIH); R01HL147155-02 (NIH)
Record Dates: First submitted 2021-01-28; First posted 2021-02-15 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-05

CONDITIONS: Bone Tumor; Cancer of Bone; Heart Diseases; Cognitive Impairment; Cognitive Decline; Chemotherapy Effect; Memory Problem
Keywords: Endoprosthesis; Metallosis; Toxicity
MeSH Terms: conditions — Bone Neoplasms; Heart Diseases; Cognitive Dysfunction; Memory Disorders | interventions — Surveys and Questionnaires; Interviews as Topic; Hematologic Tests; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected from patients and ran through a CyTOF procedure to identify immune cells within the samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoprosthesis: Patients with a endoprosthesis
  Interventions: Behavioral: Questionnaires; Behavioral: Interviews; Diagnostic Test: Blood Test; Diagnostic Test: Echocardiogram

INTERVENTIONS:
Behavioral: Questionnaires — The patient and an informant will be asked to complete a questionnaire about his or hers current and past physical thinking abilities.
Behavioral: Interviews — Cognition and memory interviews will take place with the patient.
Diagnostic Test: Blood Test — Three blood draws will occur to assess patients immune response, metal levels, and cardiac health.
Diagnostic Test: Echocardiogram — Each echocardiogram takes about 3 hours and 30 minutes. This test uses sound waves to look at your heart. The person doing the test will press on your chest with a machine to obtain the pictures. The pressure may be uncomfortable. The echocardiogram will involve an image enhancement agent infusion to obtain better images.

SUMMARY:
The purpose of this research is to investigate whether patients who previously had endoprosthesis surgery experience memory, thinking, or heart problems. It will also help determine how often these problems occur.

DETAILED DESCRIPTION:
At your first visit you will be asked to do the following:

1. Sign the consent document.
2. Patient Interview: An interview will be conducted by the study coordinator on the research team. They will ask your past surgical history, health history, medications, and your cognition.
3. Informant Interview: A close friend, spouse of relative of you will be interviewed about your day-day cognition.
4. Memory Interview: You will be evaluated on your memory and thinking skills three total times. One to determine baseline, and then repeated at one year and two years. You will answer questions that evaluate various thinking abilities such as concentration, memory, reasoning, and learning.
5. Blood Draw: You will have a blood draw three times (4.2-5 tablespoons) to determine your baseline, 1 year, and 2 year research results.

6: Echocardiogram: You will be asked to have three echocardiograms. One to determine baseline, and then repeated at one year and two years.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an endoprosthesis after extremity malignancy

Exclusion Criteria:

* Current fracture or infection around the endoprosthesis
* Patient is pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 patients to complete cardiology part of the study (questionnaires, blood test, echocardiogram).
  150 patients to complete cognitive part of the study (questionnaires, interviews, blood test).
  Patient groups may overlap.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Echo - Left Ventricular Ejection Fraction | Echo's will be taken at baseline, 1 year, and 2 years
  The echocardiogram will measure changes in LV ejection fraction as a percent.
Echo - Left Ventricular Mass | Echo's will be taken at baseline, 1 year, and 2 years
  The echocardiogram will measure changes in LV Mass in grams.
Echo - Heart Hypertrophy | Echo's will be taken at baseline, 1 year, and 2 years
  The echocardiogram will measure changes in concentric or eccentric hypertrophy in centimeters.
Cobalt Metal Levels | Cobalt level will be measured at baseline, 1 year, and 2 years
  The change in cobalt blood ion levels will be measured in ng/mL.
Chromium Metal Levels | Chromium level will be measured at baseline, 1 year, and 2 years
  The change in chromium blood ion levels will be measured in ng/mL.
Titanium Metal Levels | Titanium level will be measured at baseline, 1 year, and 2 years
  The change in titanium blood ion levels will be measured in ng/mL.

SECONDARY OUTCOMES:
Psychometrist Testing - Intelligence Score | Testing will occur at baseline, 1 year, and 2 years.
  The change in participants' intelligence will be measured using the Wechsler Adult Intelligence Scale. The scale is based of scores of 50 to 150. The higher the score the better the outcome. The average outcome will be a score of 100.
Psychometrist Testing - Memory Score | Testing will occur at baseline, 1 year, and 2 years.
  The change in participants' memory will be measured using the Wechsler Adult Memory Scale. The scale is based of scores of 50 to 150. The higher the score the better the outcome. The average outcome will be a score of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Houdek, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT04755140/ICF_000.pdf